CLINICAL TRIAL: NCT00570674
Title: A Phase I/II Trial of Abraxane in Combination With Carboplatin, Erbitux and Intensity Modulated Radiation Therapy (IMRT)for Treatment of Locally Advanced Squamous Cancer of the Head and Neck
Brief Title: Abraxane in Combination With Carboplatin, Erbitux and IMRT for Locally Advanced Squamous Cancer of the Head and Neck
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study did not continue to phase II due to the importance of HPV status as a prognostic factor to guide treatment decisions.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Roy B. Tishler, MD, Radiation Oncologist, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-069
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Results first posted 2016-12-12 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Basaloid Squamous Cell Carcinoma; Undifferentiated Carcinoma; Adenosquamous Cell Carcinoma
Keywords: SSCHN; Abraxane; IMRT
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Carcinoma; Carcinoma, Adenosquamous | interventions — Albumin-Bound Paclitaxel; Paclitaxel; Cetuximab; Carboplatin; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase I Dose Level 1: ACE-RT (Experimental): Phase I Dose Level 1 participants received Abraxane 20mg/m2 IV then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. One dose (400 mg/m2 IV) of Erbitux was given prior to start of radiation, then weekly at 250 mg/m2 IV. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  Interventions: Drug: Abraxane; Drug: Erbitux; Drug: Carboplatin; Radiation: Intensity Modulated Radiation Therapy
- Phase I Dose Level -1: AC-RT (Experimental): Phase I Dose Level -1 participants received Abraxane 20mg/m2 IV then carboplatin AUC 1.5 weekly IV during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  Interventions: Drug: Abraxane; Drug: Carboplatin; Radiation: Intensity Modulated Radiation Therapy
- Phase I Dose Level 2: AC-RT (Experimental): Phase I Dose Level 2 participants received Abraxane 30mg/m2 IV then carboplatin AUC 1.5 weekly IV during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  Interventions: Drug: Abraxane; Drug: Carboplatin; Radiation: Intensity Modulated Radiation Therapy
- Phase I Dose Level 3: AC-RT (Experimental): Phase I Dose Level 3 participants received Abraxane 40mg/m2 IV then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  Interventions: Drug: Abraxane; Drug: Carboplatin; Radiation: Intensity Modulated Radiation Therapy
- Phase I Dose Level 4: AC-RT (Experimental): Phase I Dose Level 4 participants received Abraxane 50mg/m2 IV then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  Interventions: Drug: Abraxane; Drug: Carboplatin; Radiation: Intensity Modulated Radiation Therapy

INTERVENTIONS:
Drug: Abraxane
  Other Names: paclitaxel
Drug: Erbitux
  Other Names: cetuximab
  Arms: Phase I Dose Level 1: ACE-RT
Drug: Carboplatin
  Other Names: paraplatin
Radiation: Intensity Modulated Radiation Therapy
  Other Names: IMRT

SUMMARY:
The purpose of the Phase I part of this research study is to determine the safest and most effective dose of Abraxane when given in combination with carboplatin and Erbitux during radiation therapy for head and neck cancer. The purpose of the Phase II part of this study is to determine the effects of the treatment on head and neck cancers, as well as to further study the safety of this treatment.

DETAILED DESCRIPTION:
Primary Objectives

1. Phase I-To identify the maximally tolerated dose (MTD) of Abraxane given with carboplatin plus concurrent IMRT (AC-RT)
2. Phase II-To evaluate efficacy in the phase II portion of the study by evaluating 2-year disease-free survival

Secondary Objectives

1. To evaluate the safety and tolerability
2. To estimate the overall response rate
3. To estimate 2-year overall survival
4. To evaluate functional outcome at 2 years with respect to speech, swallowing and overall quality of life (QoL), by determining mean duration of PEG-dependence and change in FACT-HN scores from baseline to 3, 6, 12 and 24 months.

STATISTICAL DESIGN:

The Phase I study followed a standard 3+3 dose escalation design. Four potential dose levels of Abraxane ultimately were under evaluation including a de-escalation dose level -1. [Note: Erbitux was originally planned to be given with carboplatin and Abraxane, but removed due to toxicity experienced at dose level 1.] The DLT observation period is the 7 weeks of treatment. The Phase I incorporated a10-patient expansion cohort to ensure that the toxicity at the MTD for AC-RT was acceptable. Planned enrollment for the Phase II study was 34 patients primarily to test whether 2-year disease-free survival was consistent with 75% rate as opposed to the null hypothesis of 53.5% based on prior research (RTOG 99-14).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven squamous cell carcinoma of th head and neck or its variants. Primary tumor sites eligible include nasopharynx, oral cavity, oropharynx, hypopharynx, larynx, or unknown primary SSCHN. Although they have squamous histology, tumors of the skin, nasal cavity and paranasal sinuses are excluded because their responsiveness to chemotherapy and radiotherapy may differ.
* Stage III or IV disease, without evidence of distant metastasis, according to the American Joint Committee on Cancer.
* Measurable disease, according to RECIST.
* Treatment-naive SSCHN, i.e. no prior chemotherapy, radiotherapy or attempted complete resection.
* < CTCAE v3.0 Grade 2 neuropathy
* 18 years of age or older
* ECOG Performance Status of 0 or 1
* No active alcohol addiction or other condition that, in the opinion of the study investigators, would interfere with the subject's ability to comply with the treatment plan.
* Lab values as outlined in the protocol
* Negative pregnancy test within 7 days of study entry

Exclusion Criteria:

* Pregnant or breast-feeding women, or women and men of childbearing potential not willing to use adequate contraception while receiving treatment and for at least 6 months thereafter.
* Symptomatic peripheral neuropathy Grade 2 or greater by CTCAE v3.0
* History of other malignancy within the previous 5 years, except for non-melanoma skin cancer, carcinoma in situ of the cervix, bladder or head and neck.
* Prior therapeutic radiation to the head and neck
* Other serious illness or medical conditions, including but not limited to: unstable cardiac disease or myocardial infarction within 6 months prior to study entry; history of significant neurologic disorder, including advanced dementia or uncontrolled seizure disorder; clinically significant uncontrolled infection; active peptic ulcer disease defined as unhealed or clinically active ulcer; hypercalcemia; active drug addiction including cocaine or intravenous drug use, defined as occuring within 6 months preceding diagnosis; chronic obstructive pulmonary disease; autoimmune disease requiring active therapy; severe psoriasis; chronic uncontrolled diarrhea.
* Patients who experienced involuntary weight loss of more than 20% of their body weight in the two months preceding study entry
* Concurrent treatment with any other anticancer therapy
* Prior therapy that targets the EGFR pathway
* Participation in an investigational drug trial within 30 days of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roy B. Tishler, MD, Principal Investigator — Dana-Farber Cancer Institute

IPD SHARING:
Plan to Share IPD: No
No plans to share individual participant data. However, cumulative results will be posted here and also published.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 29 participants were enrolled between November 2007 and August 2011.
Groups:
- Phase I Dose Level 4 Expansion Cohort: AC-RT: Phase I Dose Level 4 participants received Abraxane 50mg/m2 IV then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
  If no DLTs are observed at dose level 4 then ten additional participants (expansion cohort) will be enrolled at that dose level.
- All Phase II Participants: Participants received Abraxane according to the established recommended Phase II dose of Abraxane (50mg/m2 IV) then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
Period: Overall Study
Arm/Group | Phase I Dose Level 1: ACE-RT | Phase I Dose Level -1: AC-RT | Phase I Dose Level 2: AC-RT | Phase I Dose Level 3: AC-RT | Phase I Dose Level 4: AC-RT | Phase I Dose Level 4 Expansion Cohort: AC-RT | All Phase II Participants
Started | 6 | 3 | 4 | 3 | 3 | 10 | 0 (The study did not continue beyond phase I.)
Treated | 6 | 3 | 3 | 3 | 3 | 10 | 0
PEG Evaluable | 6 | 3 | 3 | 3 | 2 | 10 | 0
Completed | 6 | 3 | 3 | 3 | 3 | 10 | 0
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all treated patients.
Groups:
- All Phase I Participants: Participants received Abraxane according to the established dose escalation schedule 50mg/m2 IV then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. For Dose Level 1 participants, one dose (400 mg/m2 IV) of Erbitux was given prior to start of radiation, then weekly at 250 mg/m2 IV. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 60 [44 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 22
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28
Primary Tumor Site [Count of Participants; unit: Participants]
  Oral cavity | 3
  Oropharynx | 17
  Larynx | 4
  Unknown Primary | 2
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Abraxane Maximum Tolerated Dose (MTD) [Phase I]
Description: The Abraxane MTD in combination with carboplatin and concurrent IMRT is determined by the number of participants who experience a dose limiting toxicity (DLT). See subsequent primary outcome measure for the DLT definition. The MTD is defined as the highest dose at which fewer than one-third of participants experience a DLT. If no DLTs are observed then the MTD is not reached but the highest dose may then be the recommended phase II dose.
Time Frame: Adverse event assessments occurred weekly on treatment; The observation period for MTD evaluation incorporated the 7 weeks of treatment.
Population: The MTD was not reached on this trial but the recommended phase II dose was the highest dose of Abraxane evaluated.
Measure: Number; unit: mg weekly
Groups:
- All Phase I Participants: Participants received Abraxane according to the established dose escalation schedule then carboplatin AUC 1.5 IV weekly during the period of radiotherapy for a total of 7 weeks. For Dose Level 1 participants, one dose (400 mg/m2 IV) of Erbitux was given prior to start of radiation, then weekly at 250 mg/m2 IV. Intensity-modulated radiotherapy (IMRT) was delivered 5 days per week with the prescribed dose of 70 Gy to the gross tumor volume, given in 2 Gy daily fractions for a total of 35 fractions.
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 28
mg weekly | 50

2. Primary Outcome: Dose Limiting Toxicity (DLT) [Phase I]
Description: Dose limiting toxicities (DLT) were defined as treatment-related: 1) grade 3-4 non-hematological toxicity excluding untreated nausea, vomiting and diarrhea; dysphagia, esophagitis, mucositis/stomatitis, dermatitis/rash, 2) Grade 3 or greater febrile neutropenia occurring during chemoradiotherapy, 3) Grade 4 neutropenia lasting >/= 7 days and 4) Grade 3 thrombocytopenia. Grade 4 toxicities resulting in a treatment breaks > 7 days were considered DLTs.
Time Frame: Adverse event assessments occurred weekly on treatment; The observation period for DLT evaluation incorporated the 7 weeks of treatment.
Population: The analysis dataset is comprised of all treated patients in the dose escalation cohorts.While no DLTs were observed in the first 3 DL 1 patients, the cohort was expanded to 6 patients due to safety and tolerability concerns. Upon further review, it was resolved that the Abraxane dose should not be increased in the setting of concurrent Erbitux.
Measure: Number; unit: Participants with DLT
Arm/Group | Phase I Dose Level 1: ACE-RT | Phase I Dose Level -1: AC-RT | Phase I Dose Level 2: AC-RT | Phase I Dose Level 3: AC-RT | Phase I Dose Level 4: AC-RT
Number analyzed (Participants) | 6 | 3 | 3 | 3 | 3
Participants with DLT | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: 2-Year Disease-Free Survival [Phase II]
Description: Disease-free survival (DFS) is defined as the time from registration to the earlier of disease recurrence or death from any cause. Patients alive without a recurrence are censored at the date of last disease evaluation. 2-year disease-free survival is the probability of patients remaining alive and progression-free at 2-years from study entry estimated using Kaplan-Meier methods. Per RECIST 1.0 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or equivocal progression of non-target.
Time Frame: Disease assessments occurred 8-10 weeks following treatment end then every 4-6 weeks (yr 1), every 8-10 weeks (yr 2), quarterly (yr 3) and semiannually up to 2 yrs since last pt enrolled.
Population: The phase II portion planned to enroll 34 participants including the phase I expansion cohort but the study did not continue beyond phase I.
Arm/Group | All Phase II Participants
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Response Rate [Phase I]
Description: Overall response (OR) rate was defined as achieving partial response (PR) or complete response (CR) based on RECIST 1.0 criteria on treatment. Per RECIST 1.0 for target lesions, CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. To be assigned a status of CR or PR, changes in tumor measurements must be confirmed by repeat assessments performed no fewer than 4 weeks after the response criteria are first met. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions.
Time Frame: The primary re-staging assessment for response occurred 8-10 weeks following completion of treatment. Treatment duration was a mean (range) of 7.8 weeks (6.6-10.1).
Population: The analysis dataset is comprised of all treated phase I patients. Reporting within dose cohorts is not preferred given the small sample sizes.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 28
proportion of participants | .964 [.816 to .999]

5. Secondary Outcome: 2-Year Overall Survival [Phase I]
Description: 2-year overall survival is the proportion of patients alive at 2-years from study entry.
Time Frame: All patients were followed for survival for a minimum of 2 years. Median survival follow-up was 44.7 months (range 10-70) in this study cohort.
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 28
proportion of participants | .929 [.765 to .991]

6. Secondary Outcome: Duration PEG Therapy
Description: Estimated as the time from registration to the date of PEG removal.
Time Frame: Assessed until time of PEG removal which was up to 18.4 months in this study cohort.
Population: The analysis dataset is comprised of all patients with date of PEG removal (evaluable). Reporting within dose cohorts is not preferred given the small sample sizes.
Measure: Mean (Full Range); unit: months
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 27
months | 5.4 [2.4 to 18.4]

7. Secondary Outcome: Change in FACT-H&N Score From Baseline to 4 Months
Description: The FACT-H&N is a multidimensional, self-report QoL instrument specifically designed for use with head and neck cancer patients. It is comprised of 27 core items from the FACT-G (Version 4), an established survey which assesses the impact of cancer therapy in four domains: physical, social/family, emotional, and functional.
  [Cella, D, et al. JCO 1993(11)]. It is supplemented with a validated measure of 12 site specific items to assess for head and neck related symptoms. [D'Antonio L, Zimmerman G, et al. Cancer 1996 (77)] Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global QoL score (range: 0-156). Higher scores represent better QoL. The change score is calculated as post-baseline less baseline; therefore, a negative value indicates a decrease in score and correspondingly a decrease in QoL.
Time Frame: baseline and 4 months
Population: The analysis dataset is comprised of patients with evaluable data at the 2 assessment timepoints: baseline and 4 months.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 15
units on a scale | -21 [-34 to 16.2]
Statistical Analysis 1: Comparison: All Phase I Participants; Test type: Other; p < 0.01, Sign test

8. Secondary Outcome: Change in FACT-H&N Score From Baseline to 6 Months
Description: he FACT-H&N is a multidimensional, self-report QoL instrument specifically designed for use with head and neck cancer patients. It is comprised of 27 core items from the FACT-G (Version 4), an established survey which assesses the impact of cancer therapy in four domains: physical, social/family, emotional, and functional.
  [Cella, D, et al. JCO 1993(11)]. It is supplemented with a validated measure of 12 site specific items to assess for head and neck related symptoms. [D'Antonio L, Zimmerman G, et al. Cancer 1996 (77)] Each item is rated on a 0 to 4 Likert type scale, and then combined to produce subscale scores for each domain, as well as a global QoL score (range: 0-156). Higher scores represent better QoL. The change score is calculated as post-baseline less baseline; therefore, a negative value indicates a decrease in score and correspondingly a decrease in QoL.
Time Frame: Baseline and 6 months
Population: The analysis dataset is comprised of patients with evaluable data at the 2 assessment timepoints: baseline and 6 months.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 19
units on a scale | -9 [-28.4 to 13.3]
Statistical Analysis 1: Comparison: All Phase I Participants; Test type: Other; p < 0.01, Sign test

9. Secondary Outcome: Change in FACT-H&N Score From Baseline to 12 Months
Description: as for outcome 7
Time Frame: Baseline and 12 months
Population: The analysis dataset is comprised of patients with evaluable data at the 2 assessment timepoints: baseline and 12 months.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 17
units on a scale | -4.2 [-33 to 18]
Statistical Analysis 1: Comparison: All Phase I Participants; Test type: Other; p = 0.52, Sign test

10. Secondary Outcome: Change in FACT-H&N Score From Baseline to 24 Months
Description: as for outcome 7
Time Frame: Baseline and 24 months
Population: The analysis dataset is comprised of patients with evaluable data at the 2 assessment timepoints: baseline and 24 months.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | All Phase I Participants
Number analyzed (Participants) | 12
units on a scale | 4.3 [-25 to 24]
Statistical Analysis 1: Comparison: All Phase I Participants; Test type: Other; p = 0.39, Sign test

ADVERSE EVENTS:
Time Frame: Participants were assessed weekly on treatment and at weeks 4 and 8 post treatment. Treatment duration was a mean (range) of 7.8 weeks (6.6-10.1).
Description: Maximum grade toxicity by type was first calculated including adverse events with treatment-attribution of possibly, probably or definitely related to either chemotherapy or radiation therapy. Serious and Other AEs were defined as grades 3-5 and grades 1-2, respectively, per CTCAEv3.
Arm/Group | All Phase I Participants
Serious Adverse Events (participants affected / at risk) | 26/28
Other Adverse Events (participants affected / at risk) | 28/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Phase I Participants (N=28)
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Distention/bloating, abdominal (Gastrointestinal disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 17
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 18
Nausea (Gastrointestinal disorders) | 2
Salivary (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 1
Oral cavity, pain (Gastrointestinal disorders) | 3
Fatigue (General disorders) | 1
Edema head and neck (General disorders) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 8
Leukocytes (Investigations) | 1
Weight loss (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 1
Thrombosis/thrombus/embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Phase I Participants (N=28)
Hemoglobin (Blood and lymphatic system disorders) | 5
External ear, pain (Ear and labyrinth disorders) | 2
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 1
Middle ear, pain (Ear and labyrinth disorders) | 4
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 1
Keratitis (Eye disorders) | 1
Tearing (Eye disorders) | 1
Abdomen, pain (Gastrointestinal disorders) | 6
Constipation (Gastrointestinal disorders) | 23
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 19
Dry mouth (Gastrointestinal disorders) | 26
Dyspepsia (Gastrointestinal disorders) | 8
Dysphagia (Gastrointestinal disorders) | 9
Esophagitis (Gastrointestinal disorders) | 1
Fistula, Pancreas (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
GI-other (Gastrointestinal disorders) | 3
Hemorrhoids (Gastrointestinal disorders) | 1
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 9
Muco/stomatitis by exam, stomach (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 25
Oral cavity, pain (Gastrointestinal disorders) | 21
Salivary (Gastrointestinal disorders) | 21
Ulcer, duodenum (Gastrointestinal disorders) | 1
Ulcer, small bowel NOS (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 16
Edema head and neck (General disorders) | 14
Edema limb (General disorders) | 1
Edema trunk/genital (General disorders) | 1
Fatigue (General disorders) | 20
Fever w/o neutropenia (General disorders) | 5
Injection site reaction (General disorders) | 1
Pain-other (General disorders) | 4
Rigors/chills (General disorders) | 1
Fistula, Biliary Treet (Hepatobiliary disorders) | 1
Allergy-other (Immune system disorders) | 1
Infection Gr0-2 neut, lung (Infections and infestations) | 1
Infection Gr0-2 neut, oral cavity (Infections and infestations) | 3
Infection Gr0-2 neut, skin (Infections and infestations) | 2
Infection-other (Infections and infestations) | 16
Bruising (Injury, poisoning and procedural complications) | 1
Chemoradiation dermatitis (Injury, poisoning and procedural complications) | 18
Radiation dermatitis (Injury, poisoning and procedural complications) | 1
Leukocytes (Investigations) | 2
Neutrophils (Investigations) | 4
Platelets (Investigations) | 3
Weight loss (Investigations) | 7
Anorexia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 18
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Back, pain (Musculoskeletal and connective tissue disorders) | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1
Lymphedema-related fibrosis (Musculoskeletal and connective tissue disorders) | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 1
Dizziness (Nervous system disorders) | 1
Head/headache (Nervous system disorders) | 2
Neuropathy CN IX pharynx ear tongue (Nervous system disorders) | 1
Taste disturbance (Nervous system disorders) | 25
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 5
Confusion (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 5
Insomnia (Psychiatric disorders) | 3
Urinary frequency/urgency (Renal and urinary disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 1
Pleura, pain (Respiratory, thoracic and mediastinal disorders) | 1
Stenosis (incl anastomotic) pharynx (Respiratory, thoracic and mediastinal disorders) | 1
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 7
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 6
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Erythema multiforme (Skin and subcutaneous tissue disorders) | 5
Nail changes (Skin and subcutaneous tissue disorders) | 4
Pruritus/itching (Skin and subcutaneous tissue disorders) | 1
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 5
Skin breakdown/decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Skin-other (Skin and subcutaneous tissue disorders) | 2
Ulceration (Skin and subcutaneous tissue disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
The phase II portion planned to enroll 34 participants including the expansion cohort but the study did not continue beyond phase I given the importance of HPV status as a prognostic factor to guide treatment decisions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No